CLINICAL TRIAL: NCT02998307
Title: Optimal Serial Training Frequency for Attainment and Maintenance of High Quality CPR Using Real-Time Automated Performance Feedback Combined With Verbal Feedback From a CPR Instructor
Brief Title: Optimal Training Frequency for Attainment and Maintenance of High-quality CPR on a High-fidelity Manikin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Health Sciences North (Other)
Collaborators: Royal College of Physicians and Surgeons of Canada (Other); University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 16-010
Record Dates: First submitted 2016-12-13; First posted 2016-12-20 (Estimated); Last update posted 2018-03-15 (Actual); Status verified 2018-03

CONDITIONS: Simulation Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Monthly (Experimental): Receive bedside CPR training monthly
  Interventions: Procedure: CPR Training
- 3 months (Experimental): Receive bedside CPR training every 3 months
  Interventions: Procedure: CPR Training
- 6 months (Experimental): Receive bedside CPR training every 6 months
  Interventions: Procedure: CPR Training
- Control (No Intervention): No additional training and only performance evaluation after 1 year

INTERVENTIONS:
Procedure: CPR Training — Brief CPR assessment and training done during working hours with real-time performance feedback
  Arms: 3 months; 6 months; Monthly

SUMMARY:
Objectives: The primary objective is to determine the least frequent CPR training interval associated with continued performance of guideline-compliant CPR. The secondary objective is to determine whether certain physical characteristics, such as age, gender, exercise tolerance, height, and weight may be able to identify HCPs at high risk of being unable to perform high-quality CPR.

Design: Randomized trial to compare the effect of different training frequencies on long-term CPR performance.

Participants and setting: Nurses in all adult departments at Health Sciences North. Subjects will be randomly assigned to a group that undertakes short CPR assessment and training sessions either 1) every month, 2) every 3 months, 3) every 6 months, or 4) every 12 months (control group) over the course of a twelve-month period.

Analysis: The proportion of nurses in each group that is able to perform "excellent CPR" at the twelve-month time point will be determined. Excellent CPR is defined as a two-minute CPR session where 90% of compressions are performed with correct depth (50-60 mm), 90% with correct rate (100-120 /min), and 90% with full chest recoil. A subgroup analysis will also be performed where the demographic data of individuals who are unable to perform excellent CPR at the twelve-month time point regardless of intervention group are compared against those who are successful.

Conclusion: The results of our study will help determine the longest CPR training interval associated with maintenance of high-quality CPR skills to minimize training sessions required and decrease associated costs. The results will also generate hypotheses for future study about optimizing role assignments and team performance in resuscitation.

ELIGIBILITY:
Inclusion Criteria:

* Practicing nurses from multiple clinical environments (operating room, intensive care unit, emergency room, medical and surgical wards) at Health Sciences North.

Exclusion Criteria:

* Refusal to participate

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 244 (Actual)
Dates: Start 2016-04; Primary Completion 2017-12 (Actual); Study Completion 2018-01-08 (Actual)

PRIMARY OUTCOMES:
Proportion of nurses in each group able to perform "excellent CPR" after completing CPR training programs of various frequencies | 12 months
  "Excellent CPR" is a dichotomous variable achieved if 90% of compressions are performed with correct depth (50-60 mm), 90% with correct rate (100-120 /min), and 90% with full chest recoil.
  The proportion of nurses in each group able to perform "excellent CPR" after completing CPR training programs of various frequencies.

SECONDARY OUTCOMES:
Predictors of inability to perform high-quality CPR | 12 months
  Comparison of the following factors in participants able to perform "excellent CPR" and those who are not at the twelve-month time point: percentage of participants who are female or have self-declared shortness of breath when climbing two flights of stairs, and average age, height and weight.

CONTACTS AND LOCATIONS:
Locations (1):
- Health Sciences North, Greater Sudbury, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No